CLINICAL TRIAL: NCT06501313
Title: PhotobiomoduLation for pAtientS With Advanced hEart failuRe
Acronym: LASER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Laser Light Medical Innovations Ltd. (Unknown)
Responsible Party: Principal Investigator, Annamaria Kosztin MD, PhD, Principal Investigator, Semmelweis University Heart and Vascular Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SE-CVC-Laser 1.0
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: prospective, double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation with active device (Active Comparator)
  Interventions: Device: Photobiomodulation
- Control with Sham device (Sham Comparator)
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Soft laser therapy

SUMMARY:
The objective of the study is to examine the effectiveness of photobiomodulation therapy in patients with advanced-stage heart failure with reduced ejection fraction (HFrEF), who have been referred but ineligible for a heart transplantation. The primary endpoint is a 15% relative reduction in left ventricular end-systolic volume (LV ESV) as determined by echocardiography over a 12-month follow-up period. The secondary objective is to determine the change in NT-proBNP, a biomarker for heart failure, the change in heart failure symptoms based on the NYHA functional classification, the change in quality of life questionnaire (KCCQ), additional echocardiographic parameters, and the detection of changes in heart failure and fibrosis biomarkers. Additionally, the study aims to examine hospitalization due to heart failure and overall mortality.

ELIGIBILITY:
Inclusion Criteria:

Advanced-stage HFrEF patients who were ineligible for heart transplantation Patients over 18 years of age The expected lifespan exceeds 1 year Consent form

Exclusion Criteria:

Non-compliant patient Pregnant women Drug or alcohol abuse The patient is participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic response | 12 months
  At least 15% reduction of end-systolic volume

SECONDARY OUTCOMES:
Other echocardiographic response | 12 months
  strain alanysis, LVEF, EDV, ESV
Biomarker changes | 12 months
  NT-proBNP decrease
Symptomes | 12 months
  NYHA change
Qulaity of Life | 12 months
  KCCQ change
All-cause mortality or HF hospitalisation | 12 months

IPD SHARING:
Plan to Share IPD: No